CLINICAL TRIAL: NCT04732650
Title: Real World Difference After Changing Medication From Nonselective to Selective Endothelin Receptor Antagonist in Stable Eisenmenger Syndrome: Observational Study
Brief Title: Real World Difference After Changing Medication From Nonselective to Selective Endothelin Receptor Antagonist in Stable Eisenmenger Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Sung-A Chang, MD, Associate Professor, Samsung Medical Center
Other Study IDs: 2020-09-212
Record Dates: First submitted 2020-12-10; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Eisenmenger Complex
Keywords: pulmonary arterial hypertension; endothelin receptor antagonist; Eisenmenger complex
MeSH Terms: conditions — Eisenmenger Complex; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this study, the investigator will evaluate the treatment effects and safety, patient compliance of Ambrisentan in Eisenmenger syndrome in PAH patients who have been previously treated with Bosentan.

DETAILED DESCRIPTION:
Endothelin receptor antagonist is an established class of targeted therapy for pulmonary arterial hypertension (PAH). Nonselective ERA, Bosentan was the first approved ERA for PAH. Selective ERA, Ambrisentan was also approved for PAH treatment consequently. Although non-selective and selective ERA are both effective in clinical trials, there is no direct comparison for non-selective and selective ERA. Furthermore, approval study for both non-selective and selective ERA did not include the PAH associated with congenital heart disease (PAH-CHD) with significant shunt including Eisenmenger syndrome. Approval study for Ambrisentan;ARIES-1 and ARIES-2 trials also did not include the PAH-CHD In Korea, Bosentan was approved in 2003 and Ambrisentan was approved in 2009 for idiopathic PAH. Bosentan was also approved for PAH-CHD, however, Amrisentan was not because of limited data for PAH-CHD. Therefore, Bosentan was the only ERA covered by public health insurance since 2018 for PAH-CHD. Recently, Amrisentan was also approved for PAH associated with congenital heart disease including Eisenmger syndrome. And, there is a need for changing medication from double pill medication to once-daily dose medication because of patient's compliance.

PAH associated with CHD includes the group with significant shunt vs without shunt (s/p corrected state). When there is a shunt flow, change in pulmonary vascular resistance (PVR) and cardiac output can be a modulator of shunt flow, thus impact of pulmonary vasodilator on hemodynamics can be different from PAH without shunt. However, there is a limited data for changing ERA from non-selective to selective ERA. Our patients population can be interesting study group to understand the clinical response to changing between ERA because they are uniformly treated with non-selective ERA to selective ERA, Bosentan to Ambrisentan.

In this study, the investigators will evaluate the treatment effects and safety, patient compliance of Ambrisentan in Eisenmenger syndrome in PAH patients who have been previously treated with Bosentan.

ELIGIBILITY:
1. Inclusion Criteria

   * Age at least 18 years
   * Patient who was scheduled to change Ambrisentan from Bosentan (prospective arm) or who already changed to Ambrisentan from Bosentan (retrospective arm)
   * Presence of cyanosis with < 95 % arterial oxygen saturation (measured by transcutaneous pulse oximetry) or documented during exercise test (6 minute walk distance test or CPT stress test)
   * Bosentan treatment more than 3months before changing to Ambrisentan and stable medication dosage for 1 month before changing medication
   * Presence of PAH as diagnosed by invasive methods with Rp:Rs > 0.75 measured at rest or diagnosed by echocardiography with TR Vmax > 3.5m/s and bidirectional or right to left shunt.
   * One of the following diagnosis:

     i) non-corrected large congenital shunting defect at atrial, ventricular or arterial level: Partial anomalous venous return, atrial septal defect, ventricular septal defect, atrioventricular cushion defect, persistent ductus arteriosus, or a combination of these.

   ii) Surgically corrected shunting defect (diagnoses as above) with significant residual defect iii) Other diagnoses with univentricular physiology/haemodynamics.
2. Exclusion Criteria

   * pregnancy or lactation
   * women of child-bearing age who are sexually active without practicing reliable methods of contraception
   * any disease or impairment that, in the opinion of the investigator, excludes a subject from participation
   * substance abuse (alcohol, medicines, drugs)
   * acute decompensated heart failure within 7 days before the invasive procedure
   * significant anemia (Hb < 9.0 g/dl)
   * decompensated symptomatic polycythaemia
   * significant impairment of hepatic function (Child Pugh class C)
   * Significant left ventricular diseases (LV EF < 45%)
   * significant valvular diseases other than tricuspid or pulmonary regurgitation ( mitral or aortic valvular impairment more than moderate degree)
   * pericardial constriction
   * history of stroke, myocardial infarction or life-threatening arrhythmia within 6 months before screening
   * bronchopulmonary dysplasia or other chronic severe lung diseases
   * history of significant pulmonary embolism (in situ thromboembolism with optimal anticoagulation can be enrolled)
   * other relevant diseases (e.g. HIV infection)
   * trisomy 21
   * Unstable medication, recent changes in dosage regimen
   * Other medication with vascular action

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patient who was scheduled to change Ambrisentan from Bosentan (prospective arm) or who already changed to Ambrisentan from Bosentan (retrospective arm)
  * Presence of cyanosis with < 95 % arterial oxygen saturation (measured by transcutaneous pulse oximetry) or documented during exercise test (6 minute walk distance test or CPT stress test)
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-04 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of WHO FC | change from baseline to 6 months
  WHO functional class I, II, III, IV.
Changes in Borg dyspnea scale | change from baseline to 6 months
  scale 0 -10
TAPSE (TTE measure) | change from baseline to 6 months
  mm pericardial effusion(presence, absence), RA size(mm), RV strain(%)
pericardial effusion (TTE measure) | change from baseline to 6 months
  presence, or absence
RA size (TTE measure) | change from baseline to 6 months
  mm
RV strain(TTE measure) | change from baseline to 6 months
6-minute walk distances (6MWT) | change from baseline to 6 months
  m
blood pressure at rest (SBP and DBP) | change from baseline to 6 months
  mmHg

OTHER OUTCOMES:
adverse drug response | baseline, 12 week, 24 week, till 6 months if available.
  any adverse drug response

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bever CT Jr, Asofsky R. Augmented IgG anti-acetylcholine receptor response following chronic penicillamine administration. J Neuroimmunol. 1991 Dec;35(1-3):131-7. doi: 10.1016/0165-5728(91)90168-7. PMID 1955562
- [Background] Galie N, Beghetti M, Gatzoulis MA, Granton J, Berger RM, Lauer A, Chiossi E, Landzberg M; Bosentan Randomized Trial of Endothelin Antagonist Therapy-5 (BREATHE-5) Investigators. Bosentan therapy in patients with Eisenmenger syndrome: a multicenter, double-blind, randomized, placebo-controlled study. Circulation. 2006 Jul 4;114(1):48-54. doi: 10.1161/CIRCULATIONAHA.106.630715. Epub 2006 Jun 26. PMID 16801459
- [Background] Gatzoulis MA, Beghetti M, Galie N, Granton J, Berger RM, Lauer A, Chiossi E, Landzberg M; BREATHE-5 Investigators. Longer-term bosentan therapy improves functional capacity in Eisenmenger syndrome: results of the BREATHE-5 open-label extension study. Int J Cardiol. 2008 Jun 23;127(1):27-32. doi: 10.1016/j.ijcard.2007.04.078. Epub 2007 Jul 20. PMID 17658633